CLINICAL TRIAL: NCT03620084
Title: The Effects of Expiratory Muscle Strength Training (EMST) on Airway Protection and Swallowing in Chronic Dysphagia After Radiation Therapy
Brief Title: Effects of Expiratory Muscle Strength Training on Airway Protection and Swallowing in Chronic Dysphagia After Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2517; SHF/FG713S/2017 (Other Grant/Funding Number: SHF-Foundation)
Record Dates: First submitted 2018-07-09; First posted 2018-08-08 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Expiratory Muscle Strength Training (EMST) (Experimental): Participants will be taught how to use the EMST-150 device. The device has a one-way spring-loaded valve calibrated at different resistances that the user can select. The valve will open when expiratory pressure exceeds the threshold set by the user on the device. This threshold is set at 75% of the individual's maximum expiratory pressure for the session.
  Interventions: Device: Expiratory Muscle Strength Training (EMST)

INTERVENTIONS:
Device: Expiratory Muscle Strength Training (EMST) — The target home practice frequency on the EMST-150 is: 5 repetitions of forceful expiration each time, 5 times daily, 5 days a week for 8 weeks, following the training protocol used by Hutcheson et al. (2017).
  Other Names: EMST 150

SUMMARY:
Radiation therapy for head and neck cancer (HNC) is associated with the development of swallowing difficulties, or dysphagia. Dysphagia has profound negative effects on the health, nutritional status, and quality of life of HNC survivors. It also puts them at risk of developing life-threatening aspiration pneumonia. Radiation-associated dysphagia can be intractable and not responsive to conventional dysphagia therapy. HNC survivors with chronic severe dysphagia may be dependent on long-term tube feeding.

Expiratory Muscle Strength Training (EMST) is a low-cost, device-driven therapy. It has been studied as an approach to simultaneously improve cough and swallowing functions. During EMST, patients forcefully expire into a one-way spring-loaded valve to strengthen expiratory and submental musculature. The EMST-150 device is available for clinical use in Singapore. In other research studies, it has been shown to improve cough and swallowing in several populations of people with chronic dysphagia, most recently in people with chronic radiation-associated dysphagia.

The investigators propose to study the effect of EMST using the EMST-150 device on cough, airway protection, and swallowing functions of HNC survivors with radiation-associated dysphagia.

The investigators will recruit 40 participants to undergo an 8-week EMST programme, with weekly follow-up to calibrate their EMST device. It is hypothesised that EMST will improve participants' respiratory and swallowing functions. Respiratory function improvement will be shown by increased maximum expiratory pressure and improved cough airflow measures. Swallowing function improvement will be evidenced by reduced aspiration or improved ability to clear aspirated material during videofluoroscopic swallow studies. The investigators also hypothesize carryover effects on other aspects of swallowing, such as improved hyoid and laryngeal excursions, and improved laryngeal vestibule closure.

With the results of this study, the investigators aim to develop better evidence-based rehabilitation programmes for HNC survivors, and those living with chronic dysphagia.

ELIGIBILITY:
Inclusion criteria

* Chronic dysphagia involving the pharyngeal phase of swallowing for at least 6 months
* Undergone radiation therapy for head and neck cancer
* Penetration and/or aspiration seen on previous clinical videofluoroscopy swallow study (Penetration-Aspiration Scale score of 2 to 8)
* Failure to respond to traditional dysphagia therapy, as indicated by no improvement or only an improvement of 1 point on the Functional Oral Intake Scale, over a period of at least 4 sessions of conventional dysphagia therapy.

Exclusion criteria

* Current pneumothorax
* Severe trismus impeding insertion of rubber mouthpiece into the mouth (as part of treatment protocol)

Patients who have "perforated tympanic membrane", "history of spontaneous pneumothorax" and "history of collapsed lung", will be considered on a case-by-case basis, depending on the stability of their condition. Permission from their primary team doctors, or ENT for tympanic membrane issues, will be sought prior to enrolment into the study. These participants will only be deemed suitable for the study if their primary team doctors, ENT or respiratory doctors agree that they are stable or fully recovered, and that doing EMST will not worsen these conditions. For these patient groups, permission from the patients' primary team doctors, ENT or Respiratory Doctors will be obtained via email. Participants will not be enrolled if there is no written consent indicating approval for subject to be enrolled.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Maximum expiratory pressure | up to 8-week intervention
  cm H2O
Change in Penetration Aspiration Scale score | At baseline and end of 8-week intervention
  An 8-point rating scale of the severity of penetration and aspiration events

SECONDARY OUTCOMES:
Functional Oral Intake Scale | At baseline and end of 8-week intervention
  A 7-point scale looking at the normalcy of diet consistencies taken by the patient. The lowest score is 1 (No oral intake) and the maximum score is 7 (total oral intake with no restrictions).
Performance Status Scale-Head and Neck | At baseline and end of 8-week intervention
  An oral intake scale looking at the normalcy of diet consistencies taken by the patient. The scale ranges from 0 (tube-feeding) to 100 (full diet with no restrictions), in increments of 10.
MD Anderson Dysphagia Inventory | At baseline and end of 8-week intervention
  Self-reported swallowing-related quality of life
Modified Barium Swallow Impairment Profile | At baseline and end of 8-week intervention
  Seventeen components of swallowing are visually rated on video recordings of the modified barium swallow procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Shan Lee, BSc, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No